CLINICAL TRIAL: NCT06173830
Title: Comparison of the Effectiveness of Physical Therapy With Ultrasound-Guided Radiofrequency Ablation of the Genicular Nerve in Patients With Chronic Knee Osteoarthritis
Brief Title: Ultrasound-guided Radiofrequency Ablation of the Genicular Nerve Versus Physical Therapy for Chronic Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Merve Çakır, medical doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10026603
Record Dates: First submitted 2023-11-22; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Chronic Knee Osteoarthritis
Keywords: knee osteoarthritis; genicular nerve block; Ultrasound; radiofrequency; Chronic pain
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain | interventions — Radiofrequency Ablation; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided radiofrequency ablation of the genicular nerve in chronic knee osteoarthritis (Active Comparator): A total of 34 patients with chronic knee osteoarthritis meeting the criteria will undergo ultrasound-guided radiofrequency ablation of the genicular nerve.
  Interventions: Other: radiofrequency ablation
- physical therapy for chronic knee osteoarthritis (Active Comparator): Thirty-four patients with chronic knee osteoarthritis meeting the criteria will receive 10 sessions of physical therapy.
  Interventions: Other: physical therapy

INTERVENTIONS:
Other: radiofrequency ablation — 34 patients with chronic knee osteoarthritis meeting the criteria will undergo ultrasound-guided radiofrequency ablation of the genicular nerve.
  Arms: Ultrasound-guided radiofrequency ablation of the genicular nerve in chronic knee osteoarthritis
Other: physical therapy — 34 patients with chronic knee osteoarthritis meeting the criteria will undergo 10 sessions of physical therapy.
  Arms: physical therapy for chronic knee osteoarthritis

SUMMARY:
The aim of this study is to compare the effects of conventional physiotherapy methods with ultrasound-guided radiofrequency ablation of the genicular nerve on pain and functional status in patients with stage 2-3 chronic knee osteoarthritis.

DETAILED DESCRIPTION:
Patients diagnosed with Chronic Knee Osteoarthritis according to the American College of Rheumatology criteria, and with radiological osteoarthritis at Kellgren-Lawrence grades 2 and 3, within the age range of 45-70, and meeting the study criteria will be included in the study. After providing information about the procedures to be performed and potential risks to the patients, if they give their written informed consent, treatment methods will be applied to the patients. Eligible patients will be divided into two groups. In one group, Radiofrequency Ablation of the Genicular Nerve under Ultrasound Guidance will be performed, while the other group will receive physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* VAS ≥ 5
* To be aged between 45 and 70 years old
* Patients diagnosed with chronic knee osteoarthritis using the American College of Rheumatology criteria and having radiological osteoarthritis of Kellgren-Lawrence grade 2 and 3
* Cognitive functions being intact
* Being willing to participate in the study and signing the consent forms

Exclusion Criteria:

* Having received physical therapy for chronic knee osteoarthritis in the last 6 months
* Having received glucocorticoid or hyaluronic acid injections in the last 6 months
* Having taken oral glucosamine
* Undergoing knee surgery
* Having current neurological or mental disorders
* History of pacemaker usage
* Presence of local infections or sepsis
* Progressive neurological deficit
* Presence of oncological diseases
* Hemorrhagic diathesis or anticoagulation
* Uncontrolled diabetes or other serious internal comorbidities
* Allergy to medications or materials used
* Pregnancy
* Lack of cooperation
* Not willing to participate in the study.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Before treatment (initial), after 2 weeks and 12 weeks changes
  Scale. The Visual Analog Scale (VAS) is evaluated on a scale ranging from "no pain" to "worst possible pain." The value of 0 (zero) indicates "no pain," while the value of 10 (ten) indicates "the most severe pain imaginable."

SECONDARY OUTCOMES:
The Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Before treatment (initial), after 2 weeks and 12 weeks changes
  Questionnaire. The WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) test is a disease-specific, valid, and reliable measure for osteoarthritis, comprising 24 questions in three subcategories: pain, stiffness, and physical function. Each question is scored using the Likert scale as follows: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe. Scores for each section are calculated independently, and the total score ranges from 0 to 100. Higher scores indicate an increase in pain and stiffness, as well as a deterioration in physical function.
The 6-minute walk test (6MWT) | Before treatment (initial), after 2 weeks and 12 weeks changes
  The 6MWT is an assessment to measure the distance a person is capable of walking on a flat, hard surface in 6 minutes. It is a useful test to measure the response of all the bodily systems that a person uses while exercising.
EuroQol scale (EQ-5D-3L) | Before treatment (initial), after 2 weeks and 12 weeks changes
  Questionnaire. The EuroQol (EQ) scale, developed by the EuroQol Group, is a general tool for measuring overall quality of life. The EQ-5D-3L (3-level version) is a widely used scale for assessing health status. The EQ-5D-3L consists of two main components: the EQ-5D descriptive system and the EQ visual analog scale (EQ VAS).
  In the first component, the EQ-5D descriptive system, health status is evaluated in five dimensions: "Mobility, Self-Care, Usual Activities, Pain/Discomfort, Anxiety/Depression." Each dimension has three levels: "1=No problems," "2=Moderate problems," and "3=Severe problems." Combinations derived from these five dimensions create an index score to express individuals' overall health status.
  The second component is the visual analog scale (EQ VAS), where the patient self-assesses their health on a vertical visual analog scale with endpoints labeled 'Best imaginable health state=100' and 'Worst imaginable health state=0'.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital Physical Therapy and Rehabilitation Hospital, Ankara, Bilkent - Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi WJ, Hwang SJ, Song JG, Leem JG, Kang YU, Park PH, Shin JW. Radiofrequency treatment relieves chronic knee osteoarthritis pain: a double-blind randomized controlled trial. Pain. 2011 Mar;152(3):481-487. doi: 10.1016/j.pain.2010.09.029. Epub 2010 Nov 4. PMID 21055873
- [Background] McCormick ZL, Korn M, Reddy R, Marcolina A, Dayanim D, Mattie R, Cushman D, Bhave M, McCarthy RJ, Khan D, Nagpal G, Walega DR. Cooled Radiofrequency Ablation of the Genicular Nerves for Chronic Pain due to Knee Osteoarthritis: Six-Month Outcomes. Pain Med. 2017 Sep 1;18(9):1631-1641. doi: 10.1093/pm/pnx069. PMID 28431129
- [Result] Kesikburun S, Yasar E, Uran A, Adiguzel E, Yilmaz B. Ultrasound-Guided Genicular Nerve Pulsed Radiofrequency Treatment For Painful Knee Osteoarthritis: A Preliminary Report. Pain Physician. 2016 Jul;19(5):E751-9. PMID 27389118